CLINICAL TRIAL: NCT06365437
Title: A 12-Month, Randomized, Controlled, Open-Label, Dose Escalation Study Evaluating Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of an Anti-CD2 Monoclonal Antibody, TCD601(Siplizumab) Compared to Anti-thymocyte Globulin (rATG), as Induction Therapy in de Novo Renal Transplant Recipients
Brief Title: A Dose Escalation Study of TCD601 Compared to ATG in de Novo Renal Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: TCD601B101
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — siplizumab; Tacrolimus; Adrenal Cortex Hormones; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1 (Experimental): TCD601 administered with the contemporary standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Biological: TCD601; Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF)
- Arm 2 (Experimental): TCD601 administered with the contemporary standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Biological: TCD601; Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF)
- Arm 3 (Experimental): TCD601 administered with the contemporary standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Biological: TCD601; Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF)
- Arm 4 (Experimental): TCD601 administered with the contemporary standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Biological: TCD601; Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF)
- Arm 5 (Active Comparator): ATG administered with the contemporary standard of care (SoC) consisting of concentration-controlled tacrolimus (TAC) combined with mycophenolate mofetil (MMF) and corticosteroids (CS).
  Interventions: Drug: Tacrolimus (TAC); Drug: Corticosteroids (CS); Drug: Mycophenolate Mofetil (MMF); Drug: ATG

INTERVENTIONS:
Biological: TCD601 — Investigational Product
  Other Names: Siplizumab
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Drug: Tacrolimus (TAC) — Standard of Care Concomitant Immunosuppression
Drug: Corticosteroids (CS) — Standard of Care Concomitant Immunosuppression
Drug: Mycophenolate Mofetil (MMF) — Standard of Care Concomitant Immunosuppression
Drug: ATG — Standard of Care induction therapy in solid organ transplantation
  Arms: Arm 5

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of escalating doses of TCD601 when compared to rATG in de novo renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study requirements and provide written informed consent before and study assessment is performed.
* Male or female patients ≥ 18 to 70 years of age.
* Recipients of a de novo renal allograft from a heart-beating deceased, living unrelated, or non-HLA identical living related donor.
* Recipients of a kidney with a cold ischemia time (CIT) less than 30 hours.

Exclusion Criteria:

* Multiple-organ transplant recipients
* Subjects who have received a kidney allograft previously
* Recipient of a kidney from an HLA identical living related donor
* Recipient of a kidney from a donor after cardiac death
* Subjects at high immunological risk for rejection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | 12 months
Measure Peak Plasma Concentration (Cmax) over time. | 12 months
  The maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration.
Measure the Area under the plasma concentration versus time curve (AUC). | 12 months
  The AUC from time zero to the last measurable concentration sampling time.

SECONDARY OUTCOMES:
Assess changes in peripheral immunophenotype, including T-, B-, and NK-cells, via Fluorescence-activated Cell Sorter (FACS) over time. | 12 months
Measure anti-TCD601 antibodies in serum via Enzyme-linked Immunosorbent (ELISA) assay over time. | 12 months
Measure peripheral CD2-receptor occupancy following TCD601 administration Receptor Occupancy will be reported as the % of target saturation. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hryciw, MA, Study Director — ITB-Med LLC
Locations (7):
- Austria (2):
  - Innsbruck Medical University, Innsbruck
  - University of Vienna, Vienna
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
- Sweden (3):
  - Karolinska University Hospital, Stockholm, Huddinge
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Malmo